CLINICAL TRIAL: NCT04885985
Title: A Post Market Clinical Study to Evaluate the Safety and Efficacy of the Acotec Drug-coated Balloon in the Treatment of the Below-the-knee Artery
Brief Title: ACOART BTK RENEW：A Post Market Clinical Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acotec Scientific Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACOART BTK RENEW
Record Dates: First submitted 2021-05-10; First posted 2021-05-13 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DEB catheter (Experimental): Use DEB catheter to treat the stenosis or occlusion in below popliteal artery of experimental arm
  Interventions: Device: DEB catheter

INTERVENTIONS:
Device: DEB catheter — Trade name of DEB catheter: AcoArt Tulip (0.018") or AcoArt Litos (0.014")

SUMMARY:
The objective of this prospective, multi-center, single arm study is to obtain further data on the safety and performance of the Acotec Litos&Tulip Drug-coated Balloon catheters in the treatment of lesions in below-the-knee artery.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years old and ≤75 years old
* 2. Rutherford clinical category classification：3,4 or 5
* 3. Significant stenosis (≥70%) or occlusions of de-novo or restenotic lesion(s) located in below-the-knee arteries which distal bloodflow is patent.
* 4. Reference vessel diameter is between 2 mm and 4 mm
* 5. Subject has provided written informed consent prior to participation , understands the purpose of this trail and agrees to comply with all protocol-specified examinations and follow-up appointments.

Exclusion Criteria:

* 1. Plasma creatinine clearance rate <30 mL/min
* 2. Acute vessel occlusion or acute thrombosis in target lesion
* 3. Planned amputation on the target limb
* 4. Subjects confined to bed that are completely non-ambulatory.
* 5. Thrombolytic therapy or surgical procedure on the target limb within 6 weeks prior to enrollment.
* 6. Life expectancy < 5 year.
* 7. Cumulative length of 100% occluded target lesion(s)>150 mm
* 8. In-stent restenosis within the target lesion, or the distance between the target lesions and the stent was less than 20 mm
* 9. History of stroke within 90 days prior to enrollment
* 10. Known allergy to contrast agents, antiplatelet, anticoagulant, or thrombolytic therapy
* 11. Uncorrectable bleeding diathesis
* 12. The lesion of the inflow pathway cannot be identified due to the complete occlusion of the P3 segment of the popliteal artery
* 13. Pregnant or breastfeeding female subjects
* 14. Ability to cross a guidewire through target lesion
* 15. Patients who have participated in clinical trials of other medical devices or drugs during the same period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Estimated)
Dates: Start 2021-12-31 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Primary Patency | 6 month
  Primary patency rate is defined as freedom from clinically-driven target lesion revascularisation (CD-TLR) , restenosis as determined by duplex ultrasound (DUS) or digital subtraction angiography (DSA) or major target limb amputation.

SECONDARY OUTCOMES:
Major adverse event (MAE) rate | 30 days
  Defined as a composite rate of all-cause death, target limb major amputation and CD-TLR
Patency rate | 12 months,24 months,36 months,48 months ,60 months
  Defined as freedom from clinically-driven target lesion revascularisation (CD-TLR) , restenosis as determined by duplex ultrasound (DUS) or digital subtraction angiography (DSA) or major target limb amputation.
Rate of major target limb amputation | 12 months,24 months,36 months,48 months ,60 months
  A major adverse limb event is defined as above-ankle amputation of the treated limb
Rate of All-cause mortality | 12 months,24 months,36 months,48 months ,60 months
  All-cause mortality at 12, 24, 36, 48, 60 months post procedure
Rate of clinically-driven target vessel revascularization (CD-TVR) | 12 months,24 months,36 months,48 months ,60 months
  Clinically-driven target vessel revascularization (CD-TVR) at 12, 24, 36, 48, 60 months post procedure
Rate of clinically-driven target lesion revascularization (CD-TLR) | 12 months,24 months,36 months,48 months ,60 months
  Clinically-driven target lesion revascularization (CD-TLR) at 12, 24, 36, 48, 60 months post procedure
Rate of ulcer healing | 12 months,24 months,36 months,48 months ,60 months
  Ulcer healed or not; if not, improving, stagnant,worsening
Rate of distal embolization | through procedure completion
  Rate of distal embolization defined as occurrence significant distal embolization in target limb through the end of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Zhuang Baixi, Principal Investigator — Xiyuan Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Chui Yang Liu Hospital affiliated to Tsinghua University, Beijing, Beijing Municipality, China